CLINICAL TRIAL: NCT06977646
Title: Retrospective Study of the Surgical Treatment Restrictive Form of the Hypertrophic Cardiomyopathy Without of the Left Ventricular Outflow Tract Obstruction
Brief Title: Surgical Treatment of the Patients With Restrictive Phenotype of the Hypertrophic Cardiomyopathy Without LVOT Obstruction
Status: Enrolling by invitation | Type: Observational
Sponsor: Petrovsky National Research Centre of Surgery (Other)
Responsible Party: Sponsor
Other Study IDs: ApHCM-001
Record Dates: First submitted 2025-05-07; First posted 2025-05-18 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Apical Hypertrophic Cardiomyopathy
Keywords: Apical hypertrophic cardiomyopathy; Midventricular obstruction and cavity obliteration; Septal myectomy; hypertrophic cardiomyopathy; sudden cardiac death
MeSH Terms: conditions — Apical Hypertrophic Cardiomyopathy; Cardiomyopathy, Hypertrophic; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hypertrophic apical cardiomyopathy undergoing surgical interventions: Patients who underwent surgery for apical hypertrophic cardiomyopathy without significant left ventricular outflow tract obstruction. Patients with transapical surgical access will not be included in the study.
  Interventions: Procedure: Surgical transaortic left ventricular cavity remodeling in patients with apical hypertrophic cardiomyopathy without left ventricular outflow tract obstruction

INTERVENTIONS:
Procedure: Surgical transaortic left ventricular cavity remodeling in patients with apical hypertrophic cardiomyopathy without left ventricular outflow tract obstruction — The proposed intervention is a variation of classical myectomy, but unlike it, the main substrate for resection is not only the hypertrophied interventricular septum, but the abnormal papillary muscles and interpapillary trabeculae in the left ventricular cavity

SUMMARY:
Hypertrophic cardiomyopathy - is an inherited disease characterized by pronounced genetic and phenotypic heterogeneity. There are two most common anatomic variants of cardiac hypertrophy: subaortic and submitral phenotypes. Subaortic phenotype is characterized by hypertrophy of the basal parts of the heart, mainly in the interventricular septum (IVS), manifesting by a high pressure gradient in the LVOT. Submitral phenotype is characterized by localization of hypertrophic zone downward to the apex and apical phenotype is without a pressure gradient in the LVOT.

The morphology, nature of hemodynamic abnormalities not well studied in patients with apical phenotype of HCM, and surgical treatment are controversial, and for those patients with advanced stage of the HF the orthotopic heart transplantations (HTx) is usually considered.

One of the surgical techniques available for this category of patients is apical myectomy. The main goal of this intervention is increasing the left ventricular volume and improving of the LV compliance with an increase of the diastolic relaxation. Limited data of such procedures in HCM patients were already published but it still requires further investigation on larger cohort of patients.

In this study, the investigators hypothesize that along with left ventricular septal hypertrophy, a small cavity is formed in patients with submittal-apical phenotype due to an increased number of hypertrophied papillary muscles. They are displaced to the apex and tightly fixed both among themselves and to the left ventricular walls. This causes a significant reduction in diastolic volume and left ventricular relaxation capacity. The present study will analyze the experience of performing resection of hypertrophied trabeculae and mobilization of papillary muscles performed through the aorta. Throw this approach procedure can be done without the need for traumatic access and suturing in the apex of the left ventricle.

ELIGIBILITY:
Inclusion Criteria:

* Hypertrophic apical cardiomyopathy according to medical records
* Surgical left ventricular remodeling performed

Exclusion Criteria:

* LVOT gradient greater than 30 mmHg

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include all patients meeting the inclusion criteria treated in the period from 2017 to 2024 at the Petrovsky National Research Centre of Surgery and the Federal Cardiac Surgery Center in Astrakhan
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Hospital mortality after undergoing trans aortic surgical left ventricular remodeling | Assessment by medical records during the first 28 days after surgical intervention
  Binary value: of alive/dead

SECONDARY OUTCOMES:
left ventricular diastolic dysfunction | Perioperative/Periprocedural
  Diastolic left ventricular function relying on echo protocols. E/A ratio as an equation of an early transmitral flow (E wave) and a late flow with atrial contraction (A wave). An E/A ratio less than 0.75 or greater than 1.5 indicates dyastolic disfunction.
Heart Failure (NYHA) | 1 month after surgery
  Functional class of heart failure according to New York Heart Association (NYHA) Functional Classification of heart failure
Need for mechanical circulation in the postoperative period | Perioperative/Periprocedural
  Binary value: yes/no
Freedom from re-interventions after surgical left ventricular remodeling | hrough study completion, an average of 1 year
  Binary value yes/no According to available medical records for the entire follow-up period

OTHER OUTCOMES:
Search for mutations in full genomic DNA by sequencing method | through study completion, an average of 1 year
  Pathogenicity assessment of candidate genetic variants is performed according to the ACMG recommendations (2015) Will be performed on patients who have a preserved tissue sample suitable for whole genome sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Sergey L Dzemeshkevich, MD, PhD, Prof., Principal Investigator — Petrovsky National Research Centre of Surgery
Locations (1):
- Petrovsky National Research Centre of Surgery, Moscow, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided